CLINICAL TRIAL: NCT06146920
Title: Pilot Study Evaluation the Use of Serial Plasma Next-generation Sequencing (NGS) as a New Efficacy Metric to Guide Immunotherapy Treatment Discontinuation
Brief Title: Use of Serial Plasma NGS as a New Efficacy Metric to Guide Immunotherapy Treatment Discontinuation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Foundation Medicine (Industry)
Responsible Party: Principal Investigator, Meghan Mooradian, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-357
Record Dates: First submitted 2023-11-10; First posted 2023-11-27 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Melanoma; Non-small Cell Lung Cancer
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy

STUDY DESIGN:
Intervention Model Description: All consented participants with evidence of disease control / response after at least 1 year of immune checkpoint inhibition (monotherapy or in combination) with negative ctDNA will be invited to stop systemic therapy and continue with active surveillance.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Surveillance (Other): Patients with 12 month history of immune checkpoint inhibitors (ICI) with stable or partial or complete responses and negative ctDNA at pre-screening, will stop ICI therapy and begin active surveillance with blood draws and standard of care imaging for 12 months.
  Interventions: Other: Evaluation of ctDNA using the F1T after 1 year of immunotherapy

INTERVENTIONS:
Other: Evaluation of ctDNA using the F1T after 1 year of immunotherapy — Patients with evidence of disease control after at least 10months of an ICI-based therapy will initially undergo a pre-screen. In patients with successful F1CDx baseline tissue testing whole blood will be collected and evaluated for plasma ctDNA measurement. If there is detectable ctDNA during the pre-screening period, patients will be excluded from enrollment. If there is no detectable ctDNA, patients will be eligible to screen and enroll in the main study.
  If enrolled, patients will stop ICI- based treatment and continue with serial ctDNA at pre-specified timepoints. The treating physician will not be blinded to the serial ctDNA results There will be no proscriptive therapeutic measures outlined if ctDNA becomes detectable while on study.
  Other Names: Discontinue Immune Checkpoint Inhibitor

SUMMARY:
The goal of this prospective study to investigate the use of circulating tumor DNA (ctDNA) to guide end of therapy decisions in patients with melanoma or non-small-cell lung cancer.

The main question it aims to answer is:

• Do patients with metastatic melanoma or non-small-cell lung cancer, who have received at least 12 months of immune checkpoint inhibition (monotherapy or in combination) with evidence of disease response/control on imaging and have no evidence of circulating tumor DNA, have an increased 12-month disease free survival in comparison to historical controls?

DETAILED DESCRIPTION:
This is a prospective study using Simon's two stage design to investigate the use of ctDNA to guide end of therapy decisions. Approximately 39 patients with an established diagnosis of metastatic melanoma or NSCLC with evidence of disease control (SD, PR, or CR) will be enrolled in the study.

Patients that sign a pre-screening consent will have archival tumor tissue sent to Foundation Medicine for generation of the F1CDx. Patients may begin screening after 10 months of an ICI containing regimen with plan to complete at least 1 year of systemic therapy. After successful generation of F1CDx whole blood will be collected and analyzed for plasma ctDNA measurement.

Eligible patients for enrollment are ctDNA negative and have received at least 12 months but no more than 18moths of ICI. Eligible patients will be offered to consent to the main study and have standard of care imaging as well as blood draws for ctDNA assessment at screening, 1 month, 2 month, 3 months, 6 months, 9 months, and 12 month/end of study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age > 18) with unresectable, metastatic melanoma (cutaneous, acral, mucosal) or NSCLC who have evidence of disease control after at least 12 months of ICI based therapy (pembrolizumab, nivolumab, nivolumab-relatimab, ipilimumab/nivolumab, atezolizumab, ipilimumab, durvalumab, cemiplimab) with or without chemotherapy in the case of NSCLC. Any line of therapy is permitted with the exception of adjuvant therapy
* Participants must be actively receiving standard of care ICI-based therapy (ICI monotherapy or in combination)
* At time of enrollment patients must have received at least 12months (+/- 4 weeks) from the start of anti-PD-1 therapy and have not experienced a toxicity that prevented them from continuing therapy.
* Participants must have evidence of disease control (stable disease, partial response, or complete response) that is maintained on restaging CT scans or PET CT scans obtained at 12 months (+/- 4 weeks) from the start of initial ICI therapy
* Prior radiation to any site is allowed
* Available tumor tissue (archival) for baseline tissue testing with FoundationOne CDx or previous FoundationOne CDx testing results (within 2 years and prior test results must be after June 30, 2021)
* Life expectancy of greater than 3 months
* Participants with a prior malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment are eligible for this trial.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants with clinical or radiographic evidence of progressive disease in the 3 months prior to consideration of screening and enrollment
* Participants who are receiving an investigational agent (s)
* Participants who have had ICI discontinued due an immune-related adverse event.
* Patients with a history of an irAE but resumed ICI therapy and are receiving ICI at the time of screening are eligible to enroll.
* Participants on > 10mg of oral prednisone or its equivalent for treatment of ongoing immune-related toxicity.
* Participants who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia, endocrine toxicity requiring chronic supplementation
* Participants with a concurrent, active malignancy
* Participants in whom F1CDx generation fails
* Participants without available tumor tissue for F1CDx test result or prior F1CDx

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the 12month disease-free survival (DFS) in ctDNA negative patients | 12 months
  Disease-free survival is defined as the time of determination of ctDNA negativity to the earlier of progression or death. This will be measured in days.

SECONDARY OUTCOMES:
Overall survival of the ctDNA negative cohort | 12 months
  Overall survival is defined as the time of determination of ctDNA negativity to death. This will be measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Mooradian, MD, Principal Investigator — Massachusetts General Brigham
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu